CLINICAL TRIAL: NCT03648411
Title: Assessment of Drug Resistance Molecular Markers in Asymptomatic Malaria Among Migrant Workers in Myanmar
Brief Title: Drug Resistance Among Asymptomatic Infection
Status: Completed | Type: Observational
Sponsor: Department of Medical Research, Lower Myanmar (Other)
Collaborators: National Malaria Control Program, Myanmar (Other Government)
Responsible Party: Principal Investigator, Myat Htut Nyunt, Principal Investigator, Department of Medical Research, Lower Myanmar
Other Study IDs: DMR_2018-108
Record Dates: First submitted 2018-08-23; First posted 2018-08-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Drug Resistant Malaria; Asymptomatic Infections; Migrant Workers
Keywords: malaria; falciparum; vivax; Myanmar; migrant workers; asymptomatic infection; drug resistance
MeSH Terms: conditions — Asymptomatic Infections; Malaria

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — The DNA samples will be kept at -80 degree C according to the consent of the participants. The samples will be kept with code number and limited restricted for use in future research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shwegyin: Shwehyin is a Township in Bago Region. We will use the comparison between the two sentinel sites by the name of Shwegyin and Pinlebu. We will compare the prevalence of asymptomatic infection between these two sites. Then proportion of the drug resistance molecular markers will be compared.
  Interventions: Genetic: Drug resistance molecular markers
- Pinlebu: Pinlebu is a township in Sagaing Region. We will use the comparison between the two sentinel sites by the name of Shwegyin and Pinlebu. We will compare the prevalence of asymptomatic infection between these two sites. Then proportion of the drug resistance molecular markers will be compared.
  Interventions: Genetic: Drug resistance molecular markers

INTERVENTIONS:
Genetic: Drug resistance molecular markers — Proportion of the drug resistance molecular markers will be found-out and compared.

SUMMARY:
A cross-sectional study will be conducted in selected 2 sentinel sites for assessment of drug resistance falciparum and vivax among asymptomatic infection in migrant workers in Myanmar.

DETAILED DESCRIPTION:
Although malaria prevalence is decreasing in Myanmar, drug resistance threatens the malaria elimination by 2030 especially high risk persons including migrant population. Previous study indicated that asymptomatic malaria parasite carried drug resistance gene such as K13 mutant that is genetically responsible for artemisinin resistant falciparum malaria. These asymptomatic carries may be a source to spread the disease and it is very important to conduct the surveillance on drug resistance status among high vulnerable persons. Unfortunately, there is no study to assess the drug resistance molecular markers in asymptomatic malaria among migrant workers in Myanmar. Therefore, this study fulfills the gaps of knowledge on important of asymptomatic hidden infection exploring to formulate the recommendation for elimination of malaria in Myanmar.

In this study, asymptomatic infections are screened by rapid diagnostic test, microscopy and molecular methods.

ELIGIBILITY:
Inclusion Criteria:

* Age above 6 year
* Migrant population (moving from their normal residence place and working at a new place such as forest related activities, gold-mines or plantation sites for more than 3 months- 3 years)
* Both sex
* Participant who give informed-consent to participate the study

Exclusion Criteria:

* Known clinical malaria cases regardless of the species detected
* Patients with clinical symptoms of malaria at the time of examination
* Known history of malaria within 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The activity will cover the migrant population of the Shwegyin Township (Bago Region) and Pinlebu Township (Sagaing Region).
Sampling Method: Non-Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2019-01-12 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Prevalence of the asymptomatic infection among the study population | 1 week
  Number of the hidden malaria cases by RDT, microscopy or nested PCR (molecular method)
Proportion of the drug resistance molecular markers among asymptomatic infections | 3 months
  Among the asymptomatic cases, molecular markers will be analyzed (K13 and pfmdr1 copy number for falciparum and pvcrt-o, pvmdr1, pvdhps and pvdhfr gene analysis for vivax cases by Sanger Sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Myat H Nyunt, PhD, Principal Investigator — Department of Medical Research
Locations (1):
- Dr. Myat Phone Kyaw, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided